CLINICAL TRIAL: NCT02754908
Title: Effectiveness of Musical Training in the Improvement of the Neurocognitive Function and Psychological Well-being of Children Surviving Brain Tumours
Brief Title: Effectiveness of Musical Training in Children Surviving Brain Tumours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW16-023
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Brain Neoplasms; Child
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): In addition to medical follow-up, the subjects in the experimental group will receive weekly 45-minute lessons on musical training for one year (52 weeks), conducted by the Music Children Foundation. Qualified orchestral performers will provide the musical training. Training will start at the lowest level (hitting simple notes) and end at the highest level (able to play an entire song). The subjects will continue on to the next level if they successfully pass the relevant test; those who do not will be encouraged to repeat test.
  Interventions: Behavioral: musical training
- Placebo Control group (Placebo Comparator): The subjects will receive medical follow-up according to the schedule of the oncology units.
  They will receive the same amount of time and attention as those in the experimental group but not in a way designed to have any specific effect on the outcome measures. They will be invited to attend free, weekly 45-minute tutoring classes organised by the community for one year (52 weeks).
  Interventions: Behavioral: tutoring classes

INTERVENTIONS:
Behavioral: musical training — The subjects in the experimental group will receive weekly 45-minute lessons on musical training for one year (52 weeks), conducted by the Music Children Foundation.
  Arms: Experimental group
Behavioral: tutoring classes — They will be invited to attend free, weekly 45-minute tutoring classes organised by the community for one year (52 weeks).
  Arms: Placebo Control group

SUMMARY:
This study aims to examine the effects of musical training on improving the neurocognitive function and psychological well-being of children surviving brain tumours. Half of the participants will receive weekly 45-minute lessons on musical training for one year (52 weeks) while the other half are the placebo controls.

DETAILED DESCRIPTION:
Children surviving brain tumours have the highest risk of suffering neurocognitive late effects, such as impairment of intellectual development and deficits in attention and concentration, working memory, processing speed and executive function. Such effects severely affect their levels of academic achievement, psychosocial function and quality of life. Musical training is considered to have potential for treating neurocognitive impairment,mostly because the extensive brain networks engaged in musical training can induce substantial neuroplasticity changes in cortical and subcortical regions of motor, auditory and speech processing networks. A review of musical training for neuro-rehabilitation revealed that it can enhance motor recovery and neuroplasticity after stroke and improve motor deficits observed in Parkinson's disease. A growing body of evidence points to the beneficial effects of musical training on the cognitive development of children. The results of a longitudinal study on the effects of musical training on children's brain and cognitive development demonstrated that such training results in long-term enhancement of visualspatial, verbal and mathematical performance. Moreover, engaging in musical practice in childhood predicts academic performance and IQ at the university level. Thus, there appears to be some support for the effects of music lessons on intellectual development.

Nevertheless, although musical training is popular and is considered to be a beneficial intervention in the treatment of neurocognitive impairment, longitudinal studies that examine the efficacy of music-making in clinical settings are limited. Importantly, there is to date no study that examines the effects of musical training on induction of neuroplasticity in childhood cancer survivors with neurocognitive impairment. There is an imperative need for rigorous empirical scrutiny of the ability of musical training, in particular, to achieve neuroplasticity and thus promote the cognitive function and psychological well-being of children surviving brain tumours.

ELIGIBILITY:
Inclusion Criteria:

* surviving germ cell tumours of the brain
* be aged from 7 to 19 years
* be able to speak Cantonese and read Chinese
* have residual function of the upper extremities (i.e. be able to move the extremities, such as the fingers and arms, without assistance)
* have completed treatment for at least two months

Exclusion Criteria:

* have undertaken or are undertaking (at the time of the intervention) the study of a musical instrument following their cancer diagnosis
* with evidence of cancer recurrence or second malignancy in their medical records

Ages: 7 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in neurocognitive function from baseline at 12 month follow-up between intervention and control group | 12 month follow-up
  Subjects' IQ scores will be obtained at 12 months after starting the intervention using the Hong Kong Wechsler Intelligence Scales for Children (HK-WISC) for subjects younger than 16 years of age and the Wechsler Adult Intelligence Scale - Revised (WAIS-R) for those aged 16 years and older.
  In addition, the neuropsychological profile of each subject will also be examined at 12 months after starting the intervention. A comprehensive neuropsychological assessment is usually conducted on a one on-one basis with standardised procedures.

SECONDARY OUTCOMES:
neurocognitive function at baseline between intervention and control group | baseline
  Subjects' IQ scores will be obtained at baseline using the Hong Kong Wechsler Intelligence Scales for Children (HK-WISC) for subjects younger than 16 years of age and the Wechsler Adult Intelligence Scale - Revised (WAIS-R) for those aged 16 years and older.
  In addition, the neuropsychological profile of each subject will also be examined at baseline. A comprehensive neuropsychological assessment is usually conducted on a one on-one basis with standardised procedures.
self-esteem at baseline between intervention and control group | baseline
  The subjects' self-esteem will be assessed at baseline, using the Chinese version of the Rosenberg Self-Esteem Scale (RSES).
  The RSES is designed to measure the global self-esteem of children and adolescents. The scale comprises 10 items, rated using a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree), with total possible scores ranging from 10 to 40. Higher scores indicate higher levels of self-esteem. Participants will be asked to respond to the Chinese version of the RSES at baseline.
Change in self-esteem from baseline at 6 month follow-up between intervention and control group | 6 month follow-up
  The subjects' self-esteem will be assessed at 6 months after starting the intervention, using the Chinese version of the Rosenberg Self-Esteem Scale (RSES).
  The RSES is designed to measure the global self-esteem of children and adolescents. The scale comprises 10 items, rated using a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree), with total possible scores ranging from 10 to 40. Higher scores indicate higher levels of self-esteem.Participants will be asked to respond to the Chinese version of the RSES at 6 months after starting the intervention.
Change in self-esteem from baseline at 12 month follow-up between intervention and control group | 12 month follow-up
  The subjects' self-esteem will be assessed at 12 months after starting the intervention, using the Chinese version of the Rosenberg Self-Esteem Scale (RSES).
  The RSES is designed to measure the global self-esteem of children and adolescents. The scale comprises 10 items, rated using a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree), with total possible scores ranging from 10 to 40. Higher scores indicate higher levels of self-esteem.Participants will be asked to respond to the Chinese version of the RSES at 12 months after starting the intervention.
quality of life at baseline between intervention and control group | baseline
  The subjects' quality of life will be assessed at baseline, using the Chinese version of the Paediatric Quality of Life Inventory 4.0 Generic Core Scale (PedsQL 4.0). The PedsQL is designed to measure children's healthrelated quality of life. It comprises 23 items rated on a 5-point Likert scale. These items are categorised into four domains: physical functioning (eight items), emotional functioning (five items), social functioning (five items) and school functioning (five items). The total possible range of scores is from 0 to 100, with higher scores indicating better quality of life.Participants will be asked to respond to the Chinese version of the PedsQL 4.0 at baseline.
Change in quality of life from baseline at 6 month follow-up between intervention and control group | 6 month follow-up
  The subjects' quality of life will be assessed at 6 months after starting the intervention, using the Chinese version of the Paediatric Quality of Life Inventory 4.0 Generic Core Scale (PedsQL 4.0). The PedsQL is designed to measure children's healthrelated quality of life. It comprises 23 items rated on a 5-point Likert scale. These items are categorised into four domains: physical functioning (eight items), emotional functioning (five items), social functioning (five items) and school functioning (five items). The total possible range of scores is from 0 to 100, with higher scores indicating better quality of life. Participants will be asked to respond to the Chinese version of the PedsQL 4.0 at 6 months after starting the intervention.
Change in quality of life from baseline at 12 month follow-up between intervention and control group | 12 month follow-up
  The subjects' quality of life will be assessed at 12 months after starting the intervention, using the Chinese version of the Paediatric Quality of Life Inventory 4.0 Generic Core Scale (PedsQL 4.0). The PedsQL is designed to measure children's healthrelated quality of life. It comprises 23 items rated on a 5-point Likert scale. These items are categorised into four domains: physical functioning (eight items), emotional functioning (five items), social functioning (five items) and school functioning (five items). The total possible range of scores is from 0 to 100, with higher scores indicating better quality of life. Participants will be asked to respond to the Chinese version of the PedsQL 4.0 at 12 months after starting the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No